CLINICAL TRIAL: NCT04168762
Title: Ultrasound Effects on Human Motor Cortical Plasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20620
Record Dates: First submitted 2019-02-14; First posted 2019-11-19 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Healthy Participants
Keywords: Ultrasound; Neuromodulation; Transcranial Magnetic Stimulation; Transcranial Ultrasound Stimulation

STUDY DESIGN:
Intervention Model Description: Participants are randomized into two groups. Group A will receive a two part Transcranial Ultrasound Magnetic Stimulation (TUMS) on two visits and Group B will receive a one part TUMS on two visits.
Who Masked: Participant
Masking Description: Participants will be masks from the specific details of the type of TUMS stimulation they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TUMS and Sham Group (Experimental): During the subjects two visits they will receive a TUMS stimulation and a sham (placebo) stimulation at both visits.
  Interventions: Other: Transcranial Ultrasound Magnetic Stimulation
- TUMS or Sham Group (Experimental): During the subjects first of two visits they will receive either a TUMS stimulation or a sham (placebo) stimulation and at the second visit they will receive the other.
  Interventions: Other: Transcranial Ultrasound Magnetic Stimulation

INTERVENTIONS:
Other: Transcranial Ultrasound Magnetic Stimulation — Transcranial Ultrasound Magnetic Stimulation is a paradigm that allows for concurrent and concentric ultrasound stimulation with transcranial magnetic stimulation (TMS).

SUMMARY:
The purpose of this study is to test the duration and effect of single element focused ultrasound to the primary motor cortex on healthy human participants with the use of transcranial focused ultrasound and transcranial magnetic stimulation.

DETAILED DESCRIPTION:
Previous research has shown ultrasound to inhibit motor cortical excitability though it is currently not known how long these effects last. This is an important consideration if ultrasound is to be translated and advanced to clinical or therapeutic uses as this study will help to determine suitable ultrasound durations for efficacious use. The investigators will test the duration of ultrasound neuromodulation using transcranial magnetic stimulation which will elicit a recordable and quantifiable metric of motor cortical excitability in the form of a motor evoked potential.

Participants will complete 3 study visits. During the first study visit, participants will complete Magnetic Resonance Imaging and Computed Tomography scans for TUMS localization in visits 2 and 3. Each participant will undergo motor cortex thresholding prior to their study TUMS stimulation procedure. Depending on randomization, subjects may receive one or two TUMS stimulation procedures at each session.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult subject
* 18-65 years of age
* Provided informed consent

Exclusion Criteria:

* Presence of a significant medical, psychiatric, or neurologic illness
* History of loss of consciousness of more than ten minutes in the past year or loss of consciousness in a lifetime that required rehabilitation services
* Personal or family history of seizure
* Any history of stroke/transient ischemic attack (TIA) or severe traumatic brain injury
* Taking any medications that may decrease the threshold for seizure
* Pregnancy (self-reported)
* Affirmative answers to one or more questions of the provided attached safety questionnaires. These are not absolute contraindications to this study but the risk/benefit ratio will be carefully balanced by the PI
* Failure to follow laboratory or study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-01-27 (Estimated); Study Completion 2020-01-27 (Estimated)

PRIMARY OUTCOMES:
Change in Motor Evoked Potential Amplitude | baseline and immediately following the TUMS stimulation
  The effect of ultrasound will be measured by comparing MEP amplitude changes after TUMS compared to baseline. Baseline MEPs will be collected at the beginning of each session and changes in MEP amplitude will be measured directly after with TUMS.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided